

# STATISTICAL ANALYSIS PLAN

A Randomized, Controlled, Examiner-Blind Clinical Study Investigating the Effects of a Dentifrice Containing 0.454% w/w Stannous Fluoride on Gingivitis Treatment and Plaque Reduction When Used Twice Daily for 12 Weeks

Protocol Number: 300107

Phase: N/A

This document contains confidentiality statements that are not relevant for this publicly available version

Property of Haleon
Confidential
May not be used, divulged, published, or otherwise disclosed
without the consent of Haleon

Statistical Analysis Plan Template v7.0 



# **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Original Analysis Plan | 24-Jan-2024 | Not applicable (N/A) |



| Ta | ble of | f conter | nts | |
|---|---|---|---|---|
| | Docu | ment His | tory | 2 |
| | Table | of conte | nts | 3 |
| | List o | f Tables. | | 4 |
| Ab | breviat | ions | | 5 |
| 1 | Sumn | nary of K | Ley Protocol Information | 6 |
| | 1.1 | Study I | Design | 6 |
| | 1.2 | Study ( | Objectives | 10 |
| | 1.3 | Treatm | ents | 11 |
| | 1.4 | Sample | e Size Calculation | 12 |
| 2 | Plann | ed Analy | rses | 12 |
| | 2.1 | Interim | Analysis | 12 |
| | 2.2 | Final A | nalyses | 12 |
| 3 | Consi | iderations | s for Data Analyses and Data Handling Conventions | 13 |
| | 3.1 | Baselin | ne Definition | 13 |
| | 3.2 | Subgro | ups/Stratifications | 13 |
| | 3.3 | Centers | s Pools | 13 |
| | 3.4 | Timepo | oints and Visit Windows | 13 |
| 4 | Data . | Analysis. | | 13 |
| | 4.1 | 4.1 Populations for Analysis | | 14 |
| | | 4.1.1 | Subject Disposition | 14 |
| | | 4.1.2 | Protocol Deviations | 14 |
| | | 4.1.3 | Analysis Populations | 15 |
| | 4.2 | Subject | t Demographics and Other Baseline Characteristics | 16 |
| | | 4.2.1 | Demographic Characteristics | 16 |
| | | 4.2.2 | General Medical History | 16 |
| | 4.3 | | ents (Study Product, Rescue Medication, other Concomitant ies, Compliance) | 16 |
| | | 4.3.1 | Study Product Compliance and Exposure | 17 |
| | | 4.3.2 | Prior and Concomitant Medication | 17 |
| | 4.4 | Analys | is of Efficacy | 18 |
| | | 4.4.1 | Primary Efficacy Endpoint | 18 |
| | | 4.4.2 | Secondary Efficacy Endpoints | |
| | | 4.4.3 | Exploratory Efficacy Variables | |



| | 4.4.4 | Handling of Missing Values/Censoring/Discontinuations | 27 |
|---|---|---|---|
| 4.5 | Analysis | s of Safety | 28 |
| | 4.5.1 | Adverse Events and Serious Adverse Events | 28 |
| | 4.5.2 | Other Safety Variables | 28 |
| 4.6 | Analysis | s of Other Variables | 29 |
| | 4.6.1 | Repeatability of the Examiner | 29 |
| 5 Chai | nges to the | Protocol Defined Statistical Analysis Plan | |
| App | endix 1: Li | st of Data Displays | 33 |
| List of | Tables | | |
| Table 1-1 | l | Schedule of Activities | 8 |
| Table 1-2 | 2 | Study Objectives and Endpoints | 10 |
| Table 1-3 | 3 | Investigational/Study Product Supplies | 11 |
| Table 4-1 | l | Bleeding Index Scoring System | 18 |
| Table 4-2 | 2 | Modified Gingival Index Scoring System | 23 |
| Table 4-3 | 3 | Turesky Plaque Index Scoring System | 24 |
| Table 5-1 | 1 | Changes to the Protocol Defined Statistical Analysis Plan | |



# **Abbreviations**

| - 110 10 1 0 1 1 101 101 0 | |
|----------------------------|----------------------------------------------|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| BDRM | Blind Data Review Meeting |
| BI | Bleeding Index |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CS | Compound Symmetry |
| ICF | Informed Consent Form |
| LOCF | Last Observation Carried Forward |
| LS | Least Square |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MFC | Master Formulation Code |
| MGI | Modified Gingival Index |
| mITT | Modified Intent-to-Treat |
| MMRM | Mixed Model for Repeated Measures |
| NBS | Number of Bleeding Sites |
| OHT | Oral Hard Tissue |
| OST | Oral Soft Tissue |
| PP | Per-Protocol |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SE | Standard Error |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TPI | Turesky Plaque Index |
| w/w | Weight for Weight |
| WHODD | World Health Organization Drug Dictionary |



The purpose of this Statistical Analysis Plan (SAP) is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 300107 (Version 2.0, dated 10-Oct-2023).

# 1 Summary of Key Protocol Information

The purpose of this trial is to demonstrate the efficacy and safety of a dentifrice containing 0.454% stannous fluoride (SnF<sub>2</sub>), on gingivitis treatment and plaque reduction, compared to a regular fluoride dentifrice after 12 weeks twice daily brushing in a population of clinically diagnosed gingivitis without undergoing dental prophylaxis. Gingival health and plaque reduction will be evaluated using bleeding index (BI), number of bleeding sites (NBS), modified gingival index (MGI) and Turesky modification of the Quigley Hein Plaque Index (TPI).

The study will follow a randomized, controlled, single blind (examiner blind), two-treatment arm, parallel study. Study subjects will be over 18 years old, non-smokers, in good general health with clinically measurable levels of gingivitis that meet all study criteria at the Screening and Baseline visits.

Approximately 160 subjects (approximately 80 per group) will be randomized to ensure approximately 144 evaluable subjects (approximately 72 per group) complete the study.

# 1.1 Study Design

This will be a single center, controlled, single blind (examiner blind), randomized, two--treatment arm, parallel study. Study subjects will be over 18 years old, non-smokers, in good general health with clinically measurable levels of gingivitis that meet all study criteria at the Screening and Baseline visits.

Approximately 160 subjects (approximately n=80 per group) will be randomized to ensure approximately 144 evaluable subjects (approximately 72 per group) complete the study.

This study will consist of 5 study visits: Screening, Baseline, Week 3, 6 and 12. Gingivitis will be assessed using MGI (Lobene et al, 1986) and BI (Saxton and van der Ouderaa, 1989). (The NBS will be derived from BI assessment). Plaque will be assessed using TPI (Lobene et al, 1982).

All evaluable teeth (in relation to the inclusion/ exclusion general dentition criteria) will be assessed.

At the Screening visit (Visit 1), subjects will provide their written informed consent to participate in the study. Demographics, medical history, and current medications will be recorded, followed by an oral examination (oral soft tissue (OST) examination, oral hard tissue (OHT) examination, dentition exclusions, a gross gingival assessment and pocket depth assessment).





Eligible subjects will be given a washout dentifrice and toothbrush to use in between Screening and Baseline Visits. They will also be issued with a study diary to record product usage.

Within 14±3 days of Screening (Visit 1), eligible subjects will return to the site for the Baseline visit (Visit 2) with overnight plaque (subjects will be instructed to abstain from oral hygiene for 12 hours [+6 hours; -2 hours] immediately before the visit).

At the Baseline visit, subjects will undergo, in the following order, a full OST examination, gingival inflammation (MGI), gingival bleeding (BI), supra-gingival plaque (TPI). Subjects with bleeding sites % (derived from BI assessment) or TPI score outside the inclusion criteria range will be discontinued from the study at this visit. Eligible subjects will be stratified according to their sex (male or female) to ensure a balance of sex across both treatment groups and then randomized to study product. The subjects will then be instructed to brush for at least one (timed) minute at site with their assigned study product (supervised brushing) after which they will be instructed to continue using their product twice daily (morning and evening until their next visit), at least one (timed) minute each time.

After using the study dentifrice for 3, 6, and 12 weeks, subjects will return to the study site (Visits 3, 4, and 5, respectively) with overnight plaque (subjects will be instructed to abstain from overnight toothbrushing for 12 hours [+6 hours; -2 hours] immediately before each assessment visit), at approximately the same time of day as the Baseline visit. The study dentifrice and the diary will be reviewed to determine treatment compliance. Subjects will have a full OST examination and then undergo, in the following order, MGI, BI, and TPI. At Visit 5, subjects will also have a full OHT examination, return all study supplies and have a dental prophylaxis if deemed appropriate by the investigator or examiner.

At Visits 2, 3, 4, and 5, repeatability data will be generated for MGI and TPI assessments from replicate examinations on the same subject (the subject for the MGI repeat assessment and the subject for the TPI repeat assessment can be different). Depending on subject visit scheduling, every effort will be made to complete one repeatability examination for each clinical measure during each clinical assessment day, that is, at least one MGI, and one TPI repeat assessment on each assessment day. Repeatability examinations will be separated by a minimum of 10 minutes and, where possible, separated by another subject. Due to the invasive nature of the BI assessment, it is not feasible to conduct an accurate repeatability assessment for this index.

Safety and oral tolerability of the study dentifrices will be monitored over the 12-week usage period by review of TEAEs. Medical device incidents will be recorded (the medical device in this study is the manual toothbrush used to apply the study toothpastes) throughout the study.

Table 1-1 presents the schedule of activities.



Table 1-1 Schedule of Activities

| Procedure/Assessment | Screening | | Study Visits | | | |
|---|---|---|---|---|---|---|
| | Visit 1 | | Visit 2<br>Day 0<br>Baseline <sup>1</sup> | Visit 3<br>Day 21±3<br>(Week 3)¹ | Visit 4<br>Day 42±4<br>(Week 6) <sup>1</sup> | Visit 5<br>Day 84±4<br>(Week 12)¹ |
| Informed consent | X | | | | | |
| Medical history | Х | - | | | | |
| Demographics | Х | - | | | | |
| Current/prior/concomitant medication review | Х | - | Х | Х | Х | Х |
| OST Examination | Х | | Х | Х | Х | Х |
| OHT Examination | Х | - | | | | Х |
| Gross gingival assessment <sup>2</sup> | Х | - | | | | |
| Pocket Depth Assessment <sup>2</sup> | X | - | | | | |
| Review of Inclusion/exclusion Criteria | x | ays | х | | | |
| Subject eligibility | X | ±3 d | X | | | |
| Subject continuance | | days | | X | Х | X |
| Dispense toothbrush<br>washout toothpaste, and<br>washout diary <sup>3</sup> | × | Nashout period 14 days±3 days | | | | |
| Return Washout<br>Toothpaste/Toothbrush | | Vashou | Х | | | |
| Modified Gingival Index (MGI) assessment | | | X | X | X | X |
| MGI repeatability assessment <sup>4</sup> | | _ | X | X | X | X |
| Bleeding Index (BI) assessment <sup>5</sup> | | _ | X | X | X | X |
| Plaque disclosure and plaque index (TPI) assessments | | - | х | х | х | х |
| TPI repeatability assessment <sup>6</sup> | | - | Х | х | Х | Х |
| Randomization | | - | X | | | |
| Dispense study products, timer, and study diary | | <b>-</b> | Х | | | |



| Oral hygiene instruction & supervised brushing with study dentifrice <sup>7</sup> | | × | х | х | |
|---|---|---|---|---|---|
| Review diary completion | | Х | Х | Х | X |
| Collect study products,<br>assess compliance, and<br>return to subject | | | х | х | |
| Return study products (end of study) | | | | | Х |
| End of study dental prophylaxis (optional) | | | | | Х |
| Adverse events review <sup>8</sup> | Х | X | Х | Х | Х |
| Medical device incidents review | | X | Х | Х | Х |
| Study conclusion | | | | | Х |

<u>Abbreviations:</u> OST: Oral Soft Tissue, OHT: Oral Hard Tissue, MGI: Modified Gingivitis Index, BI: bleeding index; TPI: Turesky Plaque Index.

#### Footnotes:

- 1: Subjects will abstain from overnight toothbrushing for a minimum of 12hrs (+6hr, -2hr) immediately prior to the assessment visits (Visits 2, 3, 4 and 5)
- 2: In relation to the general dentition inclusion/ exclusion criteria
- 3: No instruction or supervised brushing at screening visit
- 4: Minimum one MGI repeatability assessments during each clinical assessment day; MGI repeatability assessment at Baseline visit will be conducted after the subject's eligibility has been confirmed.
- 5: NBS and bleeding sites% are derived from BI assessment
- 6: Minimum one TPI repeatability assessments during each clinical assessment day; TPI repeatability assessment at Baseline visit will be conducted after the subject's eligibility has been confirmed.
- 7: At Baseline visit, site will confirm that 2nd toothbrush has not been used before the supervised brushing
- 8: Adverse Events (AEs), Serious Adverse Events (SAEs) and medical device incidents collected immediately after subject provides consent to participate in the study by the completion of the Informed Consent Form (ICF).



# 1.2 Study Objectives

Study objectives and endpoints are defined in Table 1-2.

Table 1-2 Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| To assess the performance of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing gingivitis, as measured by NBS, after 12 weeks twice daily toothbrushing. | At Week 12: • Change from Baseline in NBS |
| Secondary Objectives | Secondary Endpoints |
| Efficacy | , |
| To evaluate the efficacy of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing gingivitis, as measured by NBS, compared to a negative control after 12 weeks twice daily toothbrushing. | At Week 12: • Change from Baseline in NBS |
| To evaluate the efficacy of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing gingivitis, as measured by NBS, compared to a negative control, after 3 and 6 weeks twice daily toothbrushing. | At Weeks 3 & 6: • Change from Baseline in NBS |
| To evaluate the efficacy of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing plaque accumulation, as measured by the TPI (overall and interproximal), compared to a negative control, after 3, 6 and 12 weeks twice daily toothbrushing. | At Weeks 3, 6 & 12: • Change from Baseline in Mean TPI (overall and interproximal) |
| To evaluate the efficacy of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing gingivitis, as measured by BI, compared to a negative control, after 3, 6 and 12 weeks twice daily toothbrushing. | At Weeks 3, 6 & 12: • Change from Baseline in BI |
| To evaluate the efficacy of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing gingivitis, as measured by MGI, compared to a negative control, after 3, 6 and 12 weeks twice daily toothbrushing. | At Weeks 3, 6 & 12: • Change from Baseline in MGI |
| Safety To assess the oral tolerability of a dentifrice containing 0.454% w/w SnF <sub>2</sub> , over 12 weeks twice daily use. | Treatment-emergent adverse events over 12 weeks |
| Exploratory Objectives | Exploratory Endpoints |
| To explore the efficacy of a dentifrice containing 0.454% w/w SnF <sub>2</sub> in reducing gingivitis, as measured by NBS, BI and MGI, compared to a negative control, after 3, 6 | At Weeks 3, 6 & 12: Change from Baseline in NBS Mean BI |



| Objectives | Endpoints |
|---|---|
| and 12 weeks twice daily toothbrushing, in | Mean MGI |
| the low and high baseline MGI subgroup: | For each MGI subgroup |
| <ul> <li>Low: MGI ≤ 2</li> <li>High: MGI &gt; 2</li> </ul> | |
| To explore the efficacy of a dentifrice | At Weeks 3, 6 & 12: |
| containing 0.454% w/w SnF <sub>2</sub> in reducing | Change from Baseline in |
| plaque accumulation, as measured by TPI, | Mean TPI (overall and interproximal) |
| compared to a negative control, after 3, 6 | For each MGI subgroup |
| and 12 weeks twice daily toothbrushing, in | |
| the low and high baseline MGI subgroup: | |
| • Low: MGI ≤ 2 | |
| <ul> <li>High: MGI &gt; 2</li> </ul> | |

This study will be considered successful if there is a statistically significant difference in NBS after 12 weeks of twice daily brushing with the SnF2 dentifrice compared to its baseline and the difference is in favor of the SnF2 dentifrice.

#### 1.3 Treatments

Table 1-3 presents the study products.

Table 1-3 Investigational/Study Product Supplies

| Product Description | Test Product | Reference Product (negative control) |
|---|---|---|
| Product Name | Parodontax Complete Protection (0.454% w/w SnF <sub>2</sub> ) | Crest Cavity Protection (0.243% w/w sodium fluoride) |
| Pack Design | Carton of 6 over-wrapped tubes | Carton of 6 over-wrapped tubes |
| Dispensing Details | One carton – baseline visit | One carton – baseline visit |
| Product Master<br>Formulation Code<br>(MFC) | (Commercial Product) | Commercial Product |
| Dose/Application | Full ribbon of dentifrice on head of toothbrush provided | Full ribbon of dentifrice on head of toothbrush provided |
| Route of Administration | Oral | Oral |
| Usage Instructions | Subjects will brush their teeth for at least one (timed) minute twice a day (morning and evening) | Subjects will brush their teeth for at least one (timed) minute twice a day (morning and evening) |
| Return Requirements | All used/unused samples to be returned | All used/unused samples to be returned |



Detailed instructions for the return of study product/study supplies for the accountability checks and subsequent destruction which will be provided by Haleon during the study in time for study close out visit.

# 1.4 Sample Size Calculation

The primary endpoint for this study is "Change from Baseline in NBS at Week 12 for the test product (containing 0.454% w/w SnF<sub>2</sub>)". There were no previous similar studies where both a non-pre-prophylaxis was used in conjunction with the same or similar active ingredient in the test product. Thus, due to the uncertainty of what would be expected in terms of change from baseline for the test product given the aforementioned parameters, treatment efficacy estimates for the secondary objective (change from baseline in BI for test dentifrice compared to change from baseline in BI for reference dentifrice) were used instead. Two sponsor clinical studies that included pre-prophylaxis (Parkinson et al, 2014 and Haleon Study 212537) were used as reference to estimate efficacy of test dentifrice (0.45% w/w SnF<sub>2</sub>) compared to reference dentifrice (negative control). In these two studies, the mean difference between the test and reference product reported a mean difference in BI of 0.07 between groups with standard deviation (SD) ranging from 0.04 to 0.128 at 12 weeks. Due to the uncertainty of what would be expected in terms of the range of mean differences when subjects do not undergo a pre-prophylaxis, a higher SD of 0.128 was used to calculate the sample size for this study.

The percent differences from control in the reference studies remained consistent ( $\sim 40\%$  - 60% in favor of the test dentifrice) in the studies mentioned above, thus an assumption was made that these numbers would not fall far from that range in this study.

Based on the assumptions outlined above, a sample size of approximately 160 subjects (approximately 80 per group) will be randomized to ensure approximately 144 evaluable subjects (approximately 72 per group) complete the study (assuming a 10% dropout rate); this will provide sufficient power (90%) to achieve statistical significance (at the 5%, two-sided level) for the key secondary outcome.

# 2 Planned Analyses

# 2.1 Interim Analysis

No interim analysis is planned.

# 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities including any external data reconciliation have been completed and database has been locked.





3. All criteria for unblinding the randomization codes have been met and the randomization codes have been distributed.

# 3 Considerations for Data Analyses and Data Handling Conventions

#### 3.1 Baseline Definition

For all endpoints, the baseline value will be the Day 0 (Visit 2) pre-brushing assessment with a non-missing value.

Unless otherwise stated, if baseline data is missing no derivation will be performed and the baseline value will be set to missing.

# 3.2 Subgroups/Stratifications

Subjects who satisfy the study selection criteria will be stratified according to their sex (male or female) and randomized to study treatment.

Exploratory subgroup analyses will be conducted to evaluate and compare NBS, mean BI, mean MGI and mean TPI (overall and interproximal) in the low ( $\leq 2$ ) and high ( $\geq 2$ ) baseline mean MGI subgroups.

#### 3.3 Centers Pools

Since this is a single center study, pooling of centers is not applicable.

#### 3.4 Timepoints and Visit Windows

The timepoints and visits for this study are defined in Table 1-1 "Schedule of Activities". Any deviation from the study schedule may be reviewed on a case-by-case basis at the Blind Data Review Meeting (BDRM) to determine whether the data should be excluded from the Per Protocol (PP) population.

# 4 Data Analysis

Data analysis will be performed by with oversight from Haleon. The statistical analysis software used will be SAS version 9.4 or higher.

Prior to database closure a BDRM will be conducted in which various aspects of the trial will be discussed and agreed.

Except as described below, all listings will be produced for all randomized subjects.



# 4.1 Populations for Analysis

## 4.1.1 Subject Disposition

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently randomized. An enrolled subject is a subject who has signed informed consent and is eligible to proceed beyond the screening visit.

The number of subjects screened, enrolled, and randomized will be presented in Table 14.1.1.

The number and percentage of screen failure subjects (subjects not randomized) with reasons why subjects are not randomized will be displayed. Percentages for screen failure subjects will be based on the total number of subjects screened.

The number and percentage of randomized subjects who complete and discontinue the study, broken down by reason for discontinuation, will be presented by study product and overall, in Table 14.1.1. The percentages will be based on the number of subjects randomized.

Table 14.1.1 will also present the number and percentage of randomized subjects in each of the defined analysis populations (as defined in Section 4.1.3) by study product and overall. Percentages will be based on the number of subjects randomized.

Subject disposition including demographic data (age, sex, race and ethnicity), screening date, study product start date/time, subject status (completer, Yes/No), study completion or withdrawal date, duration (in days) in the study (defined as [(date of completion or withdrawal – study product start date) + 1], and the primary reason for withdrawal and further details for withdrawal will be listed (Listing 16.2.1.1) by study product.

Subject disposition information will be listed for non-randomized subjects (Listing 16.2.1.2), including demographic information (age, sex race and ethnicity), enrolled (Yes/No), screening date, reason for screen failure and any further details of reason for screen failure.

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. Data will be reviewed prior to unblinding and closure of the database to ensure all important deviations are captured and categorized. Subjects with important protocol deviations liable to influence the efficacy outcomes will be excluded from the PP population. Subjects may also be identified as having important protocol deviations not leading to exclusion from the PP population.

Important deviations of the protocol procedures may include, but will not necessarily be limited to the following:

- Consent procedures
- Inclusion or exclusion criteria
- Concomitant medication/therapy



- Study procedures
- Randomization procedures
- Study drug dosing/study product administration/study product compliance
- Visit schedule/interval
- Other

The specific details of the important protocol deviations will be listed in the Protocol Deviation Management Plan, and the assessment process will be specified in the Blind Data Review Plan. Subjects with important protocol deviations will be identified at the BDRM.

The number and percentage of subjects with at least one important protocol deviation, subjects with important protocol deviations not leading to exclusion from PP population with reasons for deviations and subjects with important protocol deviations leading to exclusion from the PP population with reasons for deviations will be presented by study product and overall, for all randomized subjects (Table 14.1.2) and listed in Listing 16.2.2.1.

All protocol deviations collected on the protocol deviation case report form (CRF) will be listed in Listing 16.2.2.2. The listing will present date of deviation, type of deviation and deviation description.

#### 4.1.3 Analysis Populations

Five analysis populations are defined.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | Comprise of all randomized subjects who receive at least one dose of the study product. This population will be based on the product the subject actually received. | <ul><li>Demographics</li><li>Safety</li></ul> |
| Modified<br>Intent-To-Treat<br>(mITT) | Comprise of all randomized subjects who complete at least one use of study product and have at least one post baseline clinical performance assessment. This population will be based on the study product to which the subject was randomized. Any subject who receives a randomization number will be considered to have been randomized. | <ul><li>Demographics</li><li>Compliance</li><li>Efficacy</li></ul> |
| Per-Protocol (PP) | Comprise of all randomized subjects who do not have any protocol deviations that could confound the interpretation of analyses conducted on the mITT. This population will be based on the study product to which the subject was randomized. | Efficacy |



| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | Protocol deviations that may exclude subjects from the PP population are defined in Section 4.1.2 (Protocol Deviations) | |
| MGI Repeatability | Comprise of all subjects who have at least one repeat MGI clinical assessment at any visit. | Repeatability for MGI |
| TPI Repeatability | Comprise of all subjects who have at least one repeat TPI clinical assessment at any visit. | Repeatability for TPI |

#### NOTES:

Please refer to Appendix 1: List of Data Displays, which details the population to be used for each display being generated.

The numbers of subjects included in each of the analysis populations will be presented (Table 14.1.1). Subjects excluded from any of the analysis populations will be listed in Listing 16.2.3.1, with the reason for exclusion.

The primary population for assessment of efficacy will be the mITT population. A PP analysis will be performed on the primary endpoint only if more than 10% of mITT subjects are excluded from the PP population. A decision on whether a PP analysis will be performed will be made prior to study unblinding (release of the randomization codes).

Any repeat clinical data collected for the repeatability assessment will only be used to assess repeatability. The main assessment of efficacy will be based on the initial assessment.

# 4.2 Subject Demographics and Other Baseline Characteristics

#### 4.2.1 Demographic Characteristics

Descriptive statistics [number of subjects (n), mean, SD, median, minimum and maximum for continuous variables, frequency count (n) and percentage (%) of subjects for categorical variables] will be presented for demographic characteristics by study product and overall. These variables include age (years), sex, race, ethnicity and baseline MGI subgroup, and will be presented for the Safety population (Table 14.1.3.1) and the mITT population (Table 14.1.3.2).

Demographic information will be listed for all randomized subjects in Listing 16.2.4.1.

#### 4.2.2 General Medical History

Medical and surgical history (in the last year) including allergies or drug sensitivity will be listed in Listing 16.2.4.2, with start date and end date or ongoing at the start of study product.

# 4.3 Treatments (Study Product, Rescue Medication, other Concomitant Therapies, Compliance)

Randomization details will be listed, including the randomization number, stratification group, the planned study product, the actual study product the subject was randomized to and the randomization date (Listing 16.1.7.1).





The study product kit allocations will be listed (Listing 16.1.7.2), including kit number and study product information.

## 4.3.1 Study Product Compliance and Exposure

Compliance data will be summarized for the mITT population and will be assessed by number of brushings.

Number of brushings, brushing compliance (%), number of missed brushings and number of additional brushings will be summarized using descriptive statistics by cumulative visit and by study product. The number and percentage of subjects <80%, between 80% - 120% and >120% compliant in each study product will also be presented by cumulative visit and by study product (Table 14.2.1).

Number of brushings is defined as: [(date of Visit x – date of Visit 2) multiplied by 2 – number of missed brushings + number of additional brushings], where x = 3, 4 and 5, respectively.

Brushing compliance (%) is defined as: [100 x (Actual number of brushings / Expected number of brushings)], where expected number of brushings is defined as: <math>[(date of Visit x - date of Visit 2) multiplied by 2].

Study product compliance (number of brushings, brushing compliance [%], number of missed brushings and number of additional brushings) will be listed in Listing 16.2.5.1 for all randomized subjects by study product.

Supervised study product application (subject number, visit, date, and time of the supervised procedure) will be listed (Listing 16.2.5.2) for all randomized subjects.

#### 4.3.2 Prior and Concomitant Medication

Prior medications/treatments, including prescription and non-prescription drugs, dietary supplements and herbal remedies, taken in the last 30 days and prior to signing the informed consent form, will be documented in the CRF. The prior and concomitant medications will be coded using a validated medication dictionary, World Health Organization Drug Dictionary (WHODD).

Prior medications and prior non-drug therapies will be listed by subject, with drug name, WHODD drug synonym, reason for medication, route, dose, frequency, start date, start day relative to the study product start date, and end date and end day relative to the study product start date (Listing 16.2.4.3) for all randomized subjects. Prior medications are defined as those which stopped before the study product start date.

Concomitant medications and concomitant non-drug therapies taken during treatment will be listed similarly (Listing 16.2.4.4) for all randomized subjects with either ongoing or end date displayed. Concomitant medications are defined as medications that started or stopped on or after the study product start date or are ongoing.



Unknown dates will not be imputed. However, if the start or stop date is unknown, then it will be assumed to be concomitant medication unless the partial start date or stop date indicates differently.

# 4.4 Analysis of Efficacy

The primary population for assessment of efficacy will be the mITT population. No repeat assessment data is to be used in any efficacy analyses.

Statistical analyses of the endpoints will be performed using the change from baseline, in order to easily present direct estimates for the within-treatment mean changes from baseline (e.g. the primary endpoint).

Descriptive summary statistics will be presented for the actual and change from baseline values at each time point.

All p-values presented will be two-sided and assessed at the 5% significance level. A sequential testing strategy will be used to adjust for multiplicity for the comparison between test and reference products in the number of bleeding sites at Week 12. This will only be assessed for confirmatory evidence if the primary endpoint (change from baseline within the test product at Week 12) achieves a statistically significant reduction. There will be no further adjustments for multiplicity for any other secondary endpoints.

## 4.4.1 Primary Efficacy Endpoint

#### 4.4.1.1 Primary Efficacy Endpoint Definition

The primary endpoint for the study is the change from baseline NBS at Week 12 in the Test Product group in the mITT population.

The BI will be assessed on the facial and lingual gingival surfaces of each scorable tooth (7-7 in each arch). Three scores (according to the scale in Table 4-1 below) should be recorded buccally/labially (distal, body and mesial sites) and three scores lingually (distal, body and mesial sites). At each visit, each subject therefore has up to 168 evaluable tooth sites (i.e. 6 measurements on up to 28 scorable teeth).

Table 4-1 Bleeding Index Scoring System

| Score | Score Description |
|-------|------------------------------------------------|
| 0 | No bleeding after 30 seconds |
| 1 | Bleeding observed within 30 seconds of probing |
| 2 | Bleeding observed immediately on probing |
| 9 | Missing tooth or not qualified tooth |



The number of bleeding sites for each subject at each visit is calculated as the number of evaluable tooth sites with a BI score of either 1 or 2, to give a count between 0 and 168 sites.

Descriptive statistics (n, mean, SD, standard error [SE], median, minimum, and maximum) will be presented for the number of bleeding sites at each time point (absolute value, change from baseline and percent change from baseline) in Table 14.2.2.1.1 for all subjects in the mITT population by study product. Raw means ( $\pm$  SE) of the number of bleeding sites at each time point will be plotted by study product in Figure 14.2.2.1.5 for all subjects in the mITT population.

Additionally, the number and percentage of subjects whose number of bleeding sites has reduced (improved), remained the same or increased (worsened), respectively compared to baseline, will be presented by study product at each time point in Table 14.2.2.1.3 for the mITT population.

Individual data for the number of bleeding sites will be listed for each subject by study product group and visit in Listing 16.2.6.1 for all randomized subjects.

## 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

The following null and alternative hypotheses will be evaluated:

- H<sub>0</sub>: There is no difference in the number of bleeding sites from baseline to Week 12 in the Test Product group.
- H<sub>1</sub>: There is a difference in the number of bleeding sites at Week 12, compared to baseline in the Test Product group.

A Mixed Model for Repeated Measures (MMRM) will be used, with change from baseline in number of bleeding sites as the dependent variable, the categorical time point (Week 3, Week 6, or Week 12), treatment group (Test Product or Reference Product) and treatment group by time point interaction as fixed effects, and baseline number of bleeding sites as a covariate. Subject will be included as a repeated measure with an unstructured covariance matrix. The Kenward Roger degrees of freedom approach will be applied. If unstructured covariance matrix does not converge, the following covariance structures will be applied in order until convergence is achieved: 1) Toeplitz, 2) compound symmetry (CS).

Using the above model, the least square (LS) mean change from baseline in number of bleeding sites will be presented for the Test Product at Week 12, along with 95% CI and p-value, testing for a non-zero change from baseline (Table 14.2.2.2.1).

The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results.



# 4.4.1.3 Supportive Analyses

A PP analysis will be performed on the number of bleeding sites if there is more than a 10% difference in the number of subjects between the PP and mITT populations. A decision on whether a PP analysis will be performed will be made prior to study unblinding (release of randomization codes).

A summary of the mean number of bleeding sites at each time point will be presented for the PP population in Table 14.2.2.1.2. A summary of the number and percentage of subjects at each time point whose number of bleeding sites has improved/remained the same/worsened compared to baseline will be presented for the PP population in Table 14.2.2.1.4. Statistical analysis of the mean number of bleeding sites will be presented for the PP population in Table 14.2.2.2.2. In addition, the mean number of bleeding sites at each time point will be plotted by study product for all subjects in the PP population (Figure 14.2.2.1.6).

In order to explore the sensitivity of results to the effect of missing data, the MMRM model described in Section 4.4.1.2 will be repeated using the Last Observation Carried Forward (LOCF) approach for the mITT population (Table 14.2.2.2.3) and the PP population (Table 14.2.2.2.4).

## 4.4.2 Secondary Efficacy Endpoints

All secondary endpoint analyses will be performed on the mITT population. Other than the sequential testing strategy for comparing the change from baseline in the number of bleeding sites between products (see Section 4.4), there will be no adjustment for multiplicity performed for any other secondary endpoints detailed in this section.

#### 4.4.2.1 Change from Baseline in Number of Bleeding Sites

The number of bleeding sites for each subject at each visit is calculated using the BI score, and descriptive statistics and frequency counts will be presented for the mITT population as detailed in Section 4.4.1.1.

## 4.4.2.1.1 Statistical Hypothesis, Model and Method of Analysis

For comparisons to baseline within each treatment group, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3 and Week 6 (for the Test Product group and the Reference Product group), and at Week 12 (for the Reference Product group) respectively:

- H<sub>0</sub>: There is no difference in the number of bleeding sites from baseline.
- H<sub>1</sub>: There is a difference in the number of bleeding sites compared to baseline.

For comparisons to negative control, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6, and Week 12, respectively:

• H<sub>0</sub>: There is no difference in change from baseline in the number of bleeding sites in the Test Product group compared to the Reference Product group.





• H<sub>1</sub>: There is a difference in change from baseline in the number of bleeding sites in the Test Product group compared to the Reference Product group.

The results from the MMRM described in Section 4.4.1.2 will be used to test the above hypotheses.

The LS mean change from baseline in number of bleeding sites will be presented for each study product at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero change from baseline.

The difference in LS mean change from baseline number of bleeding sites (Test Product – Reference Product) will also be presented at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero difference (Table 14.2.2.2.1). The % adjusted mean difference will also be presented.

The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Rank Sum test (between products comparisons) and Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results.

The MMRM model will be repeated using the LOCF approach for the mITT population (Table 14.2.2.2.3) and the PP population (Table 14.2.2.2.4).

## 4.4.2.2 Change from Baseline in Bleeding Index (BI)

The BI will be assessed at each evaluable tooth site for each subject at each visit as described in Section 4.4.1.1, according to the scoring system in Table 4-1. The BI score for each subject at each visit is calculated as the sum of index values over all evaluable tooth sites, divided by the number of evaluable tooth sites. Evaluable tooth sites are those scored as 0, 1 or 2, so the BI score has a range of 0 to 2.

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) will be presented for the BI score at each time point (absolute value, change from baseline and percent change from baseline) in Table 14.2.3.1.1 for the mITT population. Raw means (± SE) of the BI score at each time point will be plotted by study product in Figure 14.2.3.1.3 for all subjects in the mITT population.

Additionally, the number and percentage of subjects whose BI score has reduced (improved), remained the same and increased (worsened), respectively compared to baseline, will be presented by study product at each time point in Table 14.2.3.1.2 for the mITT population.

Individual data for the BI assessment at each evaluable tooth site will be listed for each subject in Listing 16.2.6.2.1, and individual data for the derived BI score will be listed for each subject in Listing 16.2.6.2.2, by study product group and visit for all randomized subjects.



## 4.4.2.2.1 Statistical Hypothesis, Model and Method of Analysis

For comparisons to baseline within each treatment group, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6 and Week 12, respectively:

- H<sub>0</sub>: There is no difference in the BI score from baseline.
- H<sub>1</sub>: There is a difference in the BI score compared to baseline.

For comparisons to negative control, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6, and Week 12, respectively:

- H<sub>0</sub>: There is no difference in change from baseline in the BI score in the Test Product group compared to the Reference Product group.
- H<sub>1</sub>: There is a difference in change from baseline in the BI score in the Test Product group compared to the Reference Product group.

A MMRM will be used as described in Section 4.4.1.2, with change from baseline in BI score as the dependent variable and baseline BI score as a covariate instead of baseline number of bleeding sites.

Using the above model, the LS mean change from baseline BI score will be presented for each study product at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero change from baseline.

The difference in LS mean change from baseline BI score (Test Product – Reference Product) will also be presented at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero difference (Table 14.2.3.2.1). The % adjusted mean difference will also be presented.

The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Rank Sum test (between products comparisons) and Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results.

The MMRM model will be repeated using the LOCF approach for the mITT population (Table 14.2.3.2.2).

#### 4.4.2.3 Change from Baseline in Modified Gingival Index (MGI)

The MGI will be assessed on the facial and lingual surfaces of each scorable tooth (77 in each arch). Two scores (according to the scale in Table 4-2 below) should be recorded buccally/labially (papilla and margin) and two scores lingually (papilla and margin). The exception to this is for Tooth 15 (Universal) and Tooth 18 (Universal), where the papillae assessments (both buccal and lingual) are not scoreable and not collected. At each visit, each subject therefore has up to 108 evaluable tooth sites (i.e. 4 measurements on up to 28 scorable teeth).



#### Table 4-2 Modified Gingival Index Scoring System

#### **Score Description**

- 0 Absence of inflammation
- Mild inflammation; slight change in colour, little change in colour; little change in texture of any portion of the marginal or papillary gingival unit
- 2 Mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit
- 3 Moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit
- 4 Severe inflammation; marked redness, edema and/ or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration
- 9 Missing tooth or not qualified tooth

The MGI score for each subject at each visit is calculated as the sum of index values over all evaluable tooth sites, divided by the number of evaluable tooth sites. Evaluable tooth sites are those scored as 0, 1, 2, 3 or 4 so the MGI score has a range of 0 to 4.

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) will be presented for the MGI score at each time point (absolute value, change from baseline and percent change from baseline) in Table 14.2.4.1.1 for the mITT population. Raw means (± SE) of the MGI score at each time point will be plotted by study product in Figure 14.2.4.1.3 for all subjects in the mITT population.

Additionally, the number and percentage of subjects whose MGI score has reduced (improved), remained the same and increased (worsened), respectively compared to baseline, will be presented by study product at each time point in Table 14.2.4.1.2 for the mITT population.

Individual data for the MGI assessment at each evaluable tooth site will be listed for each subject in Listing 16.2.6.3.1, and individual data for the derived MGI score will be listed for each subject in Listing 16.2.6.3.2, by study product group and visit for all randomized subjects.

#### 4.4.2.3.1 Statistical Hypothesis, Model and Method of Analysis

For comparisons to baseline within each treatment group, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6, and Week 12, respectively:

- H<sub>0</sub>: There is no difference in the MGI score from baseline.
- H<sub>1</sub>: There is a difference in the MGI score compared to baseline.

For comparisons to negative control, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6, and Week 12, respectively:

- H<sub>0</sub>: There is no difference in change from baseline in the MGI score in the Test Product group compared to the Reference Product group.
- H<sub>1</sub>: There is a difference in change from baseline in the MGI score in the Test Product group compared to the Reference Product group.





A MMRM will be used as described in Section 4.4.1.2, with change from baseline in MGI score as the dependent variable and baseline MGI score as a covariate instead of baseline number of bleeding sites.

Using the above model, the LS mean change from baseline MGI score will be presented for each study product at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero change from baseline.

The difference in LS mean change from baseline MGI score (Test Product – Reference Product) will also be presented at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero difference (Table 14.2.4.2.1 for the mITT population). The % adjusted mean difference will also be presented.

The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Rank Sum test (between products comparisons) and Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results.

The MMRM model will be repeated using the LOCF approach for the mITT population (Table 14.2.4.2.2).

## 4.4.2.4 Change from Baseline in Turesky Plaque Index (TPI)

The TPI will be used to assess plaque on all gradable teeth meeting the inclusion/exclusion criteria (natural teeth only). The TPI will be assessed on the facial and lingual surfaces of each scorable tooth (7-7 in each arch). Three scores (according to the scale in Table 4-3 below) should be recorded buccally/labially (distal, body and mesial sites) and three scores lingually (distal, body and mesial sites). At each visit, each subject therefore has up to 168 evaluable tooth sites (i.e. 6 measurements on up to 28 scorable teeth).

Table 4-3 Turesky Plaque Index Scoring System

#### **Score Description**

- 0 No plaque
- 1 Separate flecks of plaque at the cervical margin
- 2 Thin continuous band of plaque (up to 1 mm) at the cervical margin
- 3 Band of plague wider than 1 mm but covering < 1/3 of the tooth surface
- 4 Plague covering ≥ 1/3 but < 2/3 of the tooth surface
- 5 Plaque covering ≥ 2/3 of the tooth surface
- 9 Missing tooth or not qualified tooth

The overall TPI score for each subject at each visit is calculated as the sum of index values over all evaluable tooth sites, divided by the number of evaluable tooth sites. Evaluable tooth sites are those scored as 0, 1, 2, 3, 4 or 5 so the overall TPI score has a range of 0 to 5.



The interproximal TPI score for each subject at each visit is calculated as the sum of index values over all evaluable distal and mesial tooth sites, divided by the number of evaluable distal and mesial tooth sites. Similar to the overall TPI score, the interproximal TPI score has a range of 0 to 5.

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) will be presented at each time point (absolute value, change from baseline and percent change from baseline) in Table 14.2.5.1.1 for overall TPI score and in Table 14.2.5.1.3 for interproximal TPI score for the mITT population. Raw means (± SE) at each time point will be plotted by study product in Figure 14.2.5.1.5 for overall TPI score and in Figure 14.2.5.1.6 for interproximal TPI score, for the mITT population.

Additionally, the number and percentage of subjects whose score has reduced (improved), remained the same and increased (worsened), respectively compared to baseline, will be presented by study product at each time point in Table 14.2.5.1.2 (overall TPI score) and Table 14.2.5.1.4 (interproximal TPI score) for the mITT population.

Individual data for the TPI assessment at each evaluable tooth site will be listed for each subject in Listing 16.2.6.4.1, and individual data for the derived TPI score (overall and interproximal, respectively), will be listed for each subject in Listing 16.2.6.4.2, by study product group and visit for all randomized subjects.

## 4.4.2.4.1 Statistical Hypothesis, Model and Method of Analysis

For comparisons to baseline within each treatment group, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6, and Week 12, for the overall TPI score and interproximal TPI score, respectively:

- H<sub>0</sub>: There is no difference in the TPI score from baseline.
- H<sub>1</sub>: There is a difference in the TPI score compared to baseline.

For comparisons to negative control, the following null and alternative hypotheses will be evaluated for post-baseline time points at Week 3, Week 6 and Week 12, for the overall TPI score and interproximal TPI score, respectively:

- H<sub>0</sub>: There is no difference in change from baseline the TPI score in the Test Product group compared to the Reference Product group.
- H<sub>1</sub>: There is a difference in change from baseline in the TPI score in the Test Product group

Separate MMRMs will be used as described in Section 4.4.1.2, with change from baseline in TPI score (overall and interproximal, respectively) as the dependent variable and baseline TPI score (overall and interproximal, respectively) as a covariate instead of baseline number of bleeding sites.



Using the above model, the LS mean change from baseline TPI score will be presented for each study product at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero change from baseline.

The difference in LS mean change from baseline TPI score (Test Product – Reference Product) will also be presented at each post-baseline time point with corresponding 95% CIs and p-values to test for a non-zero difference (Table 14.2.5.2.1 for overall TPI, and Table 14.2.5.2.3 for interproximal TPI). The % adjusted mean difference will also be presented.

The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Rank Sum test (between products comparisons) and Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results.

The MMRM model will be repeated using the LOCF approach for the mITT population (Table 14.2.5.2.2 for overall TPI, and Table 14.2.5.2.4 for interproximal TPI).

#### 4.4.3 Exploratory Efficacy Variables

Results between study products (mean change from baseline for Test Product versus mean change from baseline for Reference Product) at each time point will also be obtained and presented in a similar manner as in the primary objective for the low and high baseline MGI subgroups in the mITT population:

Low: MGI ≤ 2High: MGI > 2

#### 4.4.3.1 Change from Baseline in NBS

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) for the NBS will be presented as described in Section 4.4.1.1 for each baseline MGI subgroup in Table 14.2.6.1.1. Raw means (± SE) at each time point will be plotted by study product for each baseline MGI subgroup separately in Figure 14.2.6.1.2.

The change from baseline in NBS will be analyzed at Week 3, Week 6 and Week 12 for each MGI subgroup separately using the same MMRM as described in Section 4.4.2.1.1 (Table 14.2.6.2.1).

#### 4.4.3.2 Change from Baseline in BI

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) for the BI score will be presented as described in Section 4.4.2.2 for each baseline MGI subgroup in Table 14.2.7.1.1. Raw means (± SE) at each time point will be plotted by study product for each baseline MGI subgroup separately in Figure 14.2.7.1.2.



The change from baseline in BI score will be analyzed at Week 3, Week 6 and Week 12 for each MGI subgroup separately using the same MMRM as described in Section 4.4.2.2.1 (Table 14.2.7.2.1).

## 4.4.3.3 Change from Baseline in MGI

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) for the MGI score will be presented as described in Section 4.4.2.3 for each baseline MGI subgroup in Table 14.2.8.1.1. Raw means (± SE) at each time point will be plotted by study product for each baseline MGI subgroup separately in Figure 14.2.8.1.2.

The change from baseline in MGI score will be analyzed at Week 3, Week 6 and Week 12 for each MGI subgroup separately using the same MMRM as described in Section 4.4.2.3.1 (Table 14.2.8.2.1).

#### 4.4.3.4 Change from Baseline in TPI

Descriptive statistics (n, mean, SD, SE, median, minimum, and maximum) will be presented as described in Section 4.4.2.4 for each baseline MGI subgroup in Table 14.2.9.1.1 for the overall TPI score and in Table 14.2.9.1.2 for the interproximal TPI score. Raw means (± SE) at each time point will be plotted by study product for each baseline MGI subgroup separately in Figure 14.2.9.1.3 for overall TPI score and in Figure 14.2.9.1.4 for interproximal TPI score.

The change from baseline in TPI score will be analyzed at Week 3, Week 6 and Week 12 for each MGI subgroup using the same MMRM as described in Section 4.4.2.4.1 (Table 14.2.9.2.1 for overall TPI, and Table 14.2.9.2.2 for interproximal TPI).

#### 4.4.4 Handling of Missing Values/Censoring/Discontinuations

For the primary analyses, missing data will not be replaced or imputed. Subjects who withdraw from the study prematurely will be included in the statistical analyses up to the point of discontinuation. Subjects who withdraw will not be replaced. In the event that a subject has no individual BI, MGI or TPI assessments available at a given visit, the number of bleeding sites, BI score, MGI score or TPI score will also be considered as missing for that visit.

Experience in previous, similar studies suggest missing data will not be prevalent. The SAS Proc Mixed implementation of the repeated measures analysis of covariance (ANCOVA) that will be used in almost all analyses, implicitly imputes any missing data based on the non-missing observations. The basic theory on which Proc Mixed is based holds even with missing data as long as the missing data are missing at random.

An additional analysis will explore the sensitivity of results to the effect of missing data on the primary and secondary efficacy endpoints. The sensitivity analysis will use the same MMRM model, but with LOCF for missing data. Only post-baseline results may be carried forward.



# 4.5 Analysis of Safety

The safety profile of the study products will be assessed with respect to adverse events (AEs), incidents and OST/OHT abnormalities in this oral health study.

#### 4.5.1 Adverse Events and Serious Adverse Events

All AEs will be reviewed by the Clinical Research Scientist or Designee prior to database lock and unblinding, and will be coded to a system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA).

AEs will be classified as oral and non-oral on the AE page of eCRF.

Treatment emergent adverse events (TEAEs) are defined as new AEs that occur on or after the first study product use (if this date is missing, a suitable alternative will be used e.g. date of randomization). AEs with an onset date/time prior to the first study product use at baseline visit will be considered as non-treatment emergent.

The following summary tables and listings will be presented by study product group.

- Table of TEAEs by SOC and PT (Table 14.3.1.1)
- Table of TEAEs by Oral/Non-Oral and PT (Table 14.3.1.2)
- Table of treatment related TEAEs by SOC and PT (Table 14.3.1.3)
- Table of treatment related TEAEs by Oral/Non-Oral and PT (Table 14.3.1.4)
- Table of non-serious TEAEs by SOC and PT (Table 14.3.1.5) [only produced if there are more than 5 AEs]
- Table of serious TEAEs by SOC and PT (Table 14.3.1.6) [only produced if there are more than 5 serious TEAEs]
- Listing of all AEs (Listing 16.2.7.1 for all randomized subjects; Listing 16.2.7.2 for non-randomized subjects)
- Listing of deaths (Listing 14.3.2.1)
- Listing of non-fatal SAEs (Listing 14.3.2.2)
- Listing of TEAEs leading to study or product discontinuation (Listing 14.3.2.3)
- Listing of TEAEs classified as Oral (Listing 14.3.2.4)

All incidents will be listed in Listing 16.2.7.3.

In the event that there is nothing to report, a null table or listing will be produced.

#### 4.5.2 Other Safety Variables

Other safety variables are listed below:

- OST examination
- OHT examination





#### 4.5.2.1 OST Examination

This procedure will be conducted by a qualified, experienced clinical examiner. The OST examination will be accomplished by direct observation and palpation with retraction aids, as appropriate. The examination will cover the oral labial mucosa (including lips), buccal mucosa, mucogingival folds, gingival mucosa, hard palate, soft palate, tonsillar area, pharyngeal area, tongue, sublingual area, submandibular area and salivary glands.

Findings from the examination will be recorded in the CRF as either normal or abnormal, with details of any abnormalities. The results of the OST examination performed at screening will be used to determine subject eligibility. Any new OST abnormality or worsening of a pre-existing condition observed by the clinical examiner or reported by the subject after the screening examination will be recorded as an AE.

Where possible, this procedure should be conducted by a single clinical examiner.

OST will be summarized (number of subjects and percentages with abnormalities, without abnormalities, or OST not examined) by visit and study product in Table 14.3.4.1 for all subjects in the Safety Population. OST examination will be listed (Listing 16.2.8.1) for all randomized subjects.

#### 4.5.2.2 OHT Examination

This procedure should be conducted by a qualified, experienced clinical examiner. The OHT examination will be accomplished by direct observation, using retraction aids as appropriate and will identify any grossly carious lesions, signs of erosive wear, enamel irregularities, tooth fracture, gross generalized dental caries decay, decalcification and faulty restorations. The presence of any implants, fixed or removable dentures, fixed or removable orthodontic braces/bands, fixed orthodontic retainers, full crowns or veneers will be recorded. Observations will be listed as either absent or present, and conditions noted as present will be described in the CRF.

Any change observed by the clinical examiner or reported by the subject after the screening examination will be recorded as an AE. The results of the OHT examination performed at Screening will be used to determine subject eligibility.

Where possible, this procedure should be conducted by a single clinical examiner.

OHT examination will be listed (Listing 16.2.8.2) for all randomized subjects.

#### 4.6 Analysis of Other Variables

## 4.6.1 Repeatability of the Examiner

Repeat MGI and TPI assessments will be performed by the clinical examiner at Day 0 (Visit 2; Baseline), Week 3 (Visit 3), Week 6 (Visit 4) and Week 12 (Visit 5). At least 1 repeat


Statistical Analysis Plan Template v7.0




assessment should be performed for each index on each clinical assessment day, that is, at least one MGI and one TPI repeat assessment on each assessment day. 'Repeat' subjects will be selected at random from those in attendance. Different subjects can be used for repeat MGI and TPI assessments. If the same subject is selected at random for repeatability assessments at multiple visits, the pairs of observations will be considered as independent for the purposes of repeatability analysis; that is, any potential within subject correlation will be ignored.

There should be a delay of at least 10 minutes between original and repeat assessments for a given subject and ideally separated by another subject. No other procedure on the subject should be carried out between the first and the repeat assessment.

Scores from the first assessment must not be visible to the examiner/scribe when the repeat assessment is carried out.

The repeat MGI and TPI assessments will be compared to the respective original assessments (excluding any tooth surfaces assessed as missing or not qualified). The repeat assessments will not be used in any efficacy analysis.

The first and second assessments of each index will be analyzed with a Fleiss-Cohen weighted kappa coefficient ( $\kappa$ ), along with the 95% CI, to assess the intra-examiner reliability. Reliability will be deemed:

- Excellent if  $\kappa > 0.75$
- Fair to good if  $0.4 \le \kappa \le 0.75$
- Poor if  $\kappa < 0.4$

#### 4.6.1.1 MGI Repeatability

The first and repeat values of the MGI for each tooth site will be combined and cross-tabulated for the MGI Repeatability population (Table 14.2.10.1). Only subjects with both first and repeat MGI assessments available for a given tooth site at the same visit will be presented and analyzed.

#### 4.6.1.2 TPI Repeatability

The first and repeat values of the TPI for each tooth site will be combined and cross-tabulated for the TPI Repeatability population (Table 14.2.10.2). Only subjects with both first and repeat TPI assessments available for a given tooth site at the same visit will be presented and analyzed.

# 5 Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 5-1 below.



Table 5-1 Changes to the Protocol Defined Statistical Analysis Plan

| Protocol | Statistical | Analysis Plan |
|---|---|---|
| Statistical Analysis Section | Statistical Analysis Plan | Rationale for Changes |
| Section 6.8: Medication/treatments taken within 28 days of signing the informed consent form will be documented as a prior medication/treatment. Section 8.1.3: Prior medications/treatments, including prescription and non-prescription drugs, dietary supplements and herbal remedies, taken in the last 30 days and prior to signing the informed consent form, will be documented in the eCRF. | Section 4.3.2: Prior medications/treatments, including prescription and non-prescription drugs, dietary supplements and herbal remedies, taken in the last 30 days and prior to signing the informed consent form, will be documented in the CRF. | There is a discrepancy between Sections 6.8 (28 days) and 8.1.3 (30 days) of the Protocol, regarding the time frame for collection of medications/treatments prior to signing of informed consent. The intended time frame is 30 days, consistent with Protocol Section 8.1.3. |
| Section 12.1: The primary endpoint for this study is "Change from Baseline in NBS at Week 12 for the test product (containing 0.454% w/w SnF <sub>2</sub> )". There were no previous similar studies where the same active ingredient in the test product was used without pre-prophylaxis. Thus, due to the uncertainty of what would be expected in terms of change from baseline for the test product given the aforementioned parameters, treatment efficacy estimates for the key secondary objective (test dentifrice compared to the reference dentifrice) were used instead. the sample size for this study. | Section 1.4: The primary endpoint for this study is "Change from Baseline in NBS at Week 12 for the test product (containing 0.454% w/w SnF2)". There were no previous similar studies where both a non-pre-prophylaxis was used in conjunction with the same or similar active ingredient in the test product. Thus, due to the uncertainty of what would be expected in terms of change from baseline for the test product given the aforementioned parameters, treatment efficacy estimates for the secondary objective (change from baseline in BI for test dentifrice compared to change from baseline in BI for reference dentifrice) were used instead. | There is a contradicting statement in the Section 12.1 of the Protocol. The text states that the sample size is based on the key secondary objective, which is NBS, but the sample size calculation is based on Bl. For correctness, Section 1.4 of the SAP clarifies that only Bl was used for the sample size calculation. |
| Section 12.2: The Per-Protocol (PP) population will include all randomized subjects who do not have any protocol deviations. | Section 4.1.3: The PP population will comprise of all randomized subjects who do not have any protocol deviations that | For consistency with previous studies using similar endpoints, where the PP specifically focuses on mITT subjects |



| Protocol | Statistical | Analysis Plan |
|---|---|---|
| Statistical Analysis Section | Statistical Analysis Plan | Rationale for Changes |
| | could confound the interpretation of analyses conducted on the mITT. | rather than just randomized subjects. |
| Section 12.3.5: Sensitivity analyses will present results from the separate ANCOVA models using only non-missing values at each single time point. | Section 4.4.4: An additional analysis will explore the sensitivity of results to the effect of missing data on the primary and secondary efficacy endpoints. The sensitivity analysis will use the same MMRM model, but with LOCF for missing data. | For consistency with previous studies using similar endpoints, sensitivity analysis will be conducted with an MMRM using LOCF imputation, rather than separate ANCOVA models by time point using only observed values. |
| No mention of a suitable non-parametric test of the primary efficacy endpoint. | Section 4.4.1.2: The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results. | For consistency with previous studies, where Wilcoxon Signed Rank p-values were added for inclusion in the Clinical Study Report. |
| No mention of a suitable nonparametric test of within group comparisons to baseline for the secondary efficacy endpoints. | Sections 4.4.2.1.1, 4.4.2.2.1, 4.4.2.3.1 and 4.4.2.4.1: The assumption of normality and homogeneity of variance in the MMRM will be investigated. In case of violation of these assumptions, a Wilcoxon Rank Sum test (between products comparisons) and Wilcoxon Signed Rank Test (within product comparisons with baseline) will be performed to support the MMRM results. | For consistency with previous studies, where Wilcoxon Signed Rank p-values were added for inclusion in the Clinical Study Report. |



Appendix 1: List of Data Displays

| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| 14.1 Demo | graphic Data | a Summary Tables a | and Figures | | | • |
| | Table | 14.1.1 | Subject Disposition | All Screened<br>Subjects | 14.1.1 | Yes |
| | Table | 14.1.2 | Incidence of Important Protocol Deviations | All Randomized<br>Subjects | 14.1.2 | |
| | Table | 14.1.3.1 | Demographic and Baseline Characteristics | Safety<br>Population | 14.1.3.1 | |
| | Table | 14.1.3.2 | Demographic and Baseline Characteristics | mITT Population | 14.1.3.1 | Yes |
| 14.2 Effica | cy Data Sum | mary Tables and Fi | igures | • | • | • |
| | Table | 14.2.1 | Summary of Brushing Compliance | mITT Population | 14.2.1 | |
| | Table | 14.2.2.1.1 | Summary of Number of Bleeding Sites | mITT Population | 14.2.2.1.1 | Yes |
| | Table | 14.2.2.1.2 | Summary of Number of Bleeding Sites | PP Population | 14.2.2.1.1 | |
| | Table | 14.2.2.1.3 | Summary of Change in Number of Bleeding Sites | mITT Population | 14.2.2.1.3 | |
| | Table | 14.2.2.1.4 | Summary of Change in Number of Bleeding Sites | PP Population | 14.2.2.1.3 | |
| | Figure | 14.2.2.1.5 | Number of Bleeding Sites (± SE) Plot Over<br>Time by Study Product | mITT Population | 14.2.2.1.5 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Figure | 14.2.2.1.6 | Number of Bleeding Sites (± SE) Plot Over<br>Time by Study Product | PP Population | 14.2.2.1.5 | |
| | Table | 14.2.2.2.1 | Statistical Analysis of Change from Baseline in Number of Bleeding Sites | mITT Population | 14.2.2.2.1 | Yes |
| | Table | 14.2.2.2.2 | Statistical Analysis of Change from Baseline in Number of Bleeding Sites | PP Population | 14.2.2.2.1 | |
| | Table | 14.2.2.2.3 | Statistical Analysis of Change from Baseline in Number of Bleeding Sites (LOCF) | mITT Population | 14.2.2.2.1 | |
| | Table | 14.2.2.2.4 | Statistical Analysis of Change from Baseline in Number of Bleeding Sites (LOCF) | PP Population | 14.2.2.2.1 | |
| | Table | 14.2.3.1.1 | Summary of Bleeding Index (BI) | mITT Population | 14.2.2.1.1 | Yes |
| | Table | 14.2.3.1.2 | Summary of Change in Bleeding Index (BI) | mITT Population | 14.2.2.1.3 | |
| | Figure | 14.2.3.1.3 | Bleeding Index (BI) (± SE) Plot Over Time by Study Product | mITT Population | 14.2.2.1.5 | |
| | Table | 14.2.3.2.1 | Statistical Analysis of Change from Baseline in Bleeding Index (BI) | mITT Population | 14.2.2.2.1 | Yes |
| | Table | 14.2.3.2.2 | Statistical Analysis of Change from Baseline in Bleeding Index (BI) (LOCF) | mITT Population | 14.2.2.2.1 | |
| | Table | 14.2.4.1.1 | Summary of Modified Gingival Index (MGI) | mITT Population | 14.2.2.1.1 | Yes |
| | Table | 14.2.4.1.2 | Summary of Change in Modified Gingival Index (MGI) | mITT Population | 14.2.2.1.3 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Figure | 14.2.4.1.3 | Modified Gingival Index (MGI) (± SE) Plot Over<br>Time by Study Product | mITT Population | 14.2.2.1.5 | |
| | Table | 14.2.4.2.1 | Statistical Analysis of Change from Baseline in Modified Gingival Index (MGI) | mITT Population | 14.2.2.2.1 | Yes |
| | Table | 14.2.4.2.2 | Statistical Analysis of Change from Baseline in Modified Gingival Index (MGI) (LOCF) | mITT Population | 14.2.2.2.1 | |
| | Table | 14.2.5.1.1 | Summary of Overall Turesky Plaque Index (TPI) | mITT Population | 14.2.2.1.1 | Yes |
| | Table | 14.2.5.1.2 | Summary of Change in Overall Turesky<br>Plaque Index (TPI) | mITT Population | 14.2.2.1.3 | |
| | Table | 14.2.5.1.3 | Summary of Interproximal Turesky Plaque Index (TPI) | mITT Population | 14.2.2.1.1 | |
| | Table | 14.2.5.1.4 | Summary of Change in Interproximal Turesky Plaque Index (TPI) | mITT Population | 14.2.2.1.3 | |
| | Figure | 14.2.5.1.5 | Overall Turesky Plaque Index (TPI) (± SE) Plot<br>Over Time by Study Product | mITT Population | 14.2.2.1.5 | |
| | Figure | 14.2.5.1.6 | Interproximal Turesky Plaque Index (TPI) (±<br>SE) Plot Over Time by Study Product | mITT Population | 14.2.2.1.5 | |
| | Table | 14.2.5.2.1 | Statistical Analysis of Change from Baseline in<br>Overall Turesky Plaque Index (TPI) | mITT Population | 14.2.2.2.1 | Yes |
| | Table | 14.2.5.2.2 | Statistical Analysis of Change from Baseline in<br>Overall Turesky Plaque Index (TPI) (LOCF) | mITT Population | 14.2.2.2.1 | |


Statistical Analysis Plan Template v7.0




| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Table | 14.2.5.2.3 | Statistical Analysis of Change from Baseline in Interproximal Turesky Plaque Index (TPI) | mITT Population | 14.2.2.2.1 | |
| | Table | 14.2.5.2.4 | Statistical Analysis of Change from Baseline in Interproximal Turesky Plaque Index (TPI) (LOCF) | mITT Population | 14.2.2.2.1 | |
| | Table | 14.2.6.1.1 | Summary of Number of Bleeding Sites by MGI Subgroup | mITT Population | 14.2.6.1.1 | |
| | Figure | 14.2.6.1.2 | Number of Bleeding Sites (± SE) Plot Over<br>Time by Study Product and MGI Subgroup | mITT Population | 14.2.6.1.2 | |
| | Table | 14.2.6.2.1 | Statistical Analysis of Change from Baseline in Number of Bleeding Sites by MGI Subgroup | mITT Population | 14.2.6.2.1 | |
| | Table | 14.2.7.1.1 | Summary of Bleeding Index (BI) by MGI<br>Subgroup | mITT Population | 14.2.6.1.1 | |
| | Figure | 14.2.7.1.2 | Bleeding Index (BI) (± SE) Plot Over Time by Study Product and MGI Subgroup | mITT Population | 14.2.6.1.2 | |
| | Table | 14.2.7.2.1 | Statistical Analysis of Change from Baseline in Bleeding Index (BI) by MGI Subgroup | mITT Population | 14.2.6.2.1 | |
| | Table | 14.2.8.1.1 | Summary of Modified Gingival Index (MGI) by MGI Subgroup | mITT Population | 14.2.6.1.1 | |
| | Figure | 14.2.8.1.2 | Modified Gingival Index (MGI) (± SE) Plot Over Time by Study Product and MGI Subgroup | mITT Population | 14.2.6.1.2 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Table | 14.2.8.2.1 | Statistical Analysis of Change from Baseline in<br>Modified Gingival Index (MGI) by MGI<br>Subgroup | mITT Population | 14.2.6.2.1 | |
| | Table | 14.2.9.1.1 | Summary of Overall Turesky Plaque Index (TPI) by MGI Subgroup | mITT Population | 14.2.6.1.1 | |
| | Table | 14.2.9.1.2 | Summary of Interproximal Turesky Plaque Index (TPI) by MGI Subgroup | mITT Population | 14.2.6.1.1 | |
| | Figure | 14.2.9.1.3 | Overall Turesky Plaque Index (TPI) (± SE) Plot<br>Over Time by Study Product and MGI<br>Subgroup | mITT Population | 14.2.6.1.2 | |
| | Figure | 14.2.9.1.4 | Interproximal Turesky Plaque Index (TPI) (±<br>SE) Plot Over Time by Study Product and MGI<br>Subgroup | mITT Population | 14.2.6.1.2 | |
| | Table | 14.2.9.2.1 | Statistical Analysis of Change from Baseline in<br>Overall Turesky Plaque Index (TPI) by MGI<br>Subgroup | mITT Population | 14.2.6.2.1 | |
| | Table | 14.2.9.2.2 | Statistical Analysis of Change from Baseline in<br>Interproximal Turesky Plaque Index (TPI) by<br>MGI Subgroup | mITT Population | 14.2.6.2.1 | |
| | Table | 14.2.10.1 | Intra-Examiner Repeatability Analysis of<br>Modified Gingival Index (MGI) | MGI<br>Repeatability<br>Population | 14.2.10.1 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Table | 14.2.10.2 | Intra-Examiner Repeatability Analysis of Turesky Plaque Index (TPI) | TPI Repeatability Population | 14.2.10.2 | |
| 14.3 Safety | Data Summa | ary Tables and Figures | | | | |
| 14.3.1 Displ | ays of Advers | se Events | | | | |
| | Table | 14.3.1.1 | Treatment Emergent Adverse Events by<br>System Organ Class and Preferred Term | Safety<br>Population | 14.3.1.1 | Yes |
| | Table | 14.3.1.2 | Treatment Emergent Adverse Events by Oral/Non-Oral and Preferred Term | Safety<br>Population | 14.3.1.2 | |
| | Table | 14.3.1.3 | Treatment Related Treatment Emergent<br>Adverse Events by System Organ Class and<br>Preferred Term | Safety<br>Population | 14.3.1.1 | |
| | Table | 14.3.1.4 | Treatment Related Treatment Emergent<br>Adverse Events by Oral/Non-Oral and<br>Preferred Term | Safety<br>Population | 14.3.1.2 | |
| | Table | 14.3.1.5 | Non-Serious Treatment Emergent Adverse<br>Events by System Organ Class and Preferred<br>Term | Safety<br>Population | 14.3.1.1 | |
| | Table | 14.3.1.6 | Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term | Safety<br>Population | 14.3.1.1 | |
| 14.3.2 Listin | ngs of Deaths | , Other Serious and Sig | gnificant Adverse Events | | | |
| | Listing | 14.3.2.1 | Deaths | All Randomized<br>Subjects | 16.2.7.1 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Listing | 14.3.2.2 | Non-Fatal Serious Adverse Events | All Randomized Subjects | 16.2.7.1 | |
| | Listing | 14.3.2.3 | Treatment Emergent Adverse Events Leading to Study or Product Discontinuation | All Randomized<br>Subjects | 16.2.7.1 | |
| | Listing | 14.3.2.4 | Treatment Emergent Adverse Events<br>Classified as Oral | All Randomized Subjects | 16.2.7.1 | |
| 14.3.3 Narra | tives of Deat | hs, Other Serious and | Certain Other Significant Adverse Events | | | |
| | NA | | | | | |
| 14.3.4 Other | Observation | s Related to Safety an | d Abnormal Laboratory Values | | | |
| | Table | 14.3.4.1 | Summary of Oral Soft Tissue Examination | Safety<br>Population | 14.3.4.1 | |
| APPENDIX | | | | | | |
| 16.1.6 Listin | g of Subjects | Receiving Test Drug(s | s)/Investigational Product(s) from Specific Batches | s, where more than o | one batch was used | |
| | NA | | | | | |
| 16.1.7 Rand | omization Sc | heme and Codes (Sub | ject identification and treatment assigned) | | | |
| | Listing | 16.1.7.1 | Randomization Information | All Randomized<br>Subjects | 16.1.7.1 | |
| | Listing | 16.1.7.2 | Kit List Allocation | All Randomized<br>Subjects | 16.1.7.2 | |
| 16.1.9 Docu | mentation of | Statistical Methods | | | | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Raw<br>output | 16.1.9.1.1 | Statistical Analysis of Change from Baseline in<br>Number of Bleeding Sites (Reference: Table<br>14.2.2.2.1) | mITT Population | SAS Output | Yes |
| | Raw<br>output | 16.1.9.1.2 | Statistical Analysis of Change from Baseline in<br>Number of Bleeding Sites (Reference: Table<br>14.2.2.2.2) | PP Population | SAS Output | |
| | Raw<br>output | 16.1.9.1.3 | Statistical Analysis of Change from Baseline in<br>Number of Bleeding Sites (LOCF) (Reference:<br>Table 14.2.2.2.3) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.1.4 | Statistical Analysis of Change from Baseline in<br>Number of Bleeding Sites (LOCF) (Reference:<br>Table 14.2.2.2.4) | PP Population | SAS Output | |
| | Raw<br>output | 16.1.9.2.1 | Statistical Analysis of Change from Baseline in Bleeding Index (BI) (Reference: Table 14.2.3.2.1) | mITT Population | SAS Output | Yes |
| | Raw<br>output | 16.1.9.2.2 | Statistical Analysis of Change from Baseline in Bleeding Index (BI) (LOCF) (Reference: Table 14.2.3.2.2) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.3.1 | Statistical Analysis of Change from Baseline in Modified Gingival Index (MGI) (Reference: Table 14.2.4.2.1) | mITT Population | SAS Output | Yes |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Raw<br>output | 16.1.9.3.2 | Statistical Analysis of Change from Baseline in<br>Modified Gingival Index (MGI) (LOCF)<br>(Reference: Table 14.2.4.2.2) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.4.1 | Statistical Analysis of Change from Baseline in<br>Overall Turesky Plaque Index (TPI)<br>(Reference: Table 14.2.5.2.1) | mITT Population | SAS Output | Yes |
| | Raw<br>output | 16.1.9.4.2 | Statistical Analysis of Change from Baseline in<br>Overall Turesky Plaque Index (TPI) (LOCF)<br>(Reference: Table 14.2.5.2.2) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.4.3 | Statistical Analysis of Change from Baseline in<br>Overall Turesky Plaque Index (TPI) by MGI<br>Subgroup (Reference: Table 14.2.2.4.5) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.4.4 | Statistical Analysis of Change from Baseline in<br>Interproximal Turesky Plaque Index (TPI)<br>(Reference: Table 14.2.5.2.3) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.5 | Statistical Analysis of Change from Baseline in<br>Number of Bleeding Sites by MGI Subgroup<br>(Reference: Table 14.2.6.2.1) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.6 | Statistical Analysis of Change from Baseline in<br>Bleeding Index (BI) by MGI Subgroup<br>(Reference: Table 14.2.7.2.1) | mITT Population | SAS Output | |



| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Raw<br>output | 16.1.9.7 | Statistical Analysis of Change from Baseline in<br>Modified Gingival Index (MGI) by MGI<br>Subgroup (Reference: Table 14.2.8.2.1) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.8.1 | Statistical Analysis of Change from Baseline in Interproximal Turesky Plaque Index (TPI) (Reference: Table 14.2.9.2.1) | mITT Population | SAS Output | |
| | Raw<br>output | 16.1.9.8.2 | Statistical Analysis of Change from Baseline in Interproximal Turesky Plaque Index (TPI) by MGI Subgroup (Reference: Table 14.2.9.2.2) | mITT Population | SAS Output | |
| 16.2 Subject | Data Listing | s | | | | |
| 16.2.1 Disco | ntinued Subj | ects | | | | |
| | Listing | 16.2.1.1 | Subject Disposition | All Randomized<br>Subjects | 16.2.1.1 | |
| | Listing | 16.2.1.2 | Subject Disposition | Non-<br>Randomized<br>Subjects | 16.2.1.2 | |
| 16.2.2 Proto | col Deviation | S | | | | |
| | Listing | 16.2.2.1 | Important Protocol Deviations | All Randomized<br>Subjects | 16.2.2.1 | |
| | Listing | 16.2.2.2 | All Protocol Deviations | All Randomized<br>Subjects | 16.2.2.2 | |
| 16.2.3 Patier | nts Excluded | from the Efficacy Anal | ysis | | | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Listing | 16.2.3.1 | Exclusions from Analysis Populations | All Randomized<br>Subjects | 16.2.3.1 | |
| 16.2.4 Dem | nographic Dat | а | | | | |
| | Listing | 16.2.4.1 | Demographic and Baseline Characteristics | All Randomized<br>Subjects | 16.2.4.1 | |
| | Listing | 16.2.4.2 | Medical History and Current Medical Conditions | All Randomized<br>Subjects | 16.2.4.2 | |
| | Listing | 16.2.4.3 | Prior Medications | All Randomized<br>Subjects | 16.2.4.3 | |
| | Listing | 16.2.4.4 | Concomitant Medications and Concomitant Non-Drug Therapies | All Randomized<br>Subjects | 16.2.4.4 | |
| 16.2.5 Com | pliance and/o | or Drug Concentration | Data (if available) | | | |
| | Listing | 16.2.5.1 | Brushing Compliance | All Randomized<br>Subjects | 16.2.5.1 | |
| | Listing | 16.2.5.2 | Supervised Brushing | All Randomized<br>Subjects | 16.2.5.2 | |
| 16.2.6 Indiv | idual Efficacy | / Response Data | | · | | - |
| | Listing | 16.2.6.1 | Number of Bleeding Sites | All Randomized<br>Subjects | 16.2.6.1 | |
| | Listing | 16.2.6.2.1 | Bleeding Index (BI) Individual Scores | All Randomized<br>Subjects | 16.2.6.2.1 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Listing | 16.2.6.2.2 | Bleeding Index (BI) Derived Scores | All Randomized<br>Subjects | 16.2.6.2.2 | |
| | Listing | 16.2.6.3.1 | Modified Gingival Index (MGI) Individual Scores | All Randomized<br>Subjects | 16.2.6.3.1 | |
| | Listing | 16.2.6.3.2 | Modified Gingival Index (MGI) Derived Scores | All Randomized<br>Subjects | 16.2.6.3.2 | |
| | Listing | 16.2.6.4.1 | Turesky Plaque Index (TPI) Individual Scores | All Randomized<br>Subjects | 16.2.6.4.1 | |
| | Listing | 16.2.6.4.2 | Turesky Plaque Index (TPI) Derived Scores | All Randomized<br>Subjects | 16.2.6.4.2 | |
| 16.2.7 Adv | erse Event Li | istings | | | | |
| | Listing | 16.2.7.1 | All Adverse Events | All Randomized<br>Subjects | 16.2.7.1 | |
| | Listing | 16.2.7.2 | All Adverse Events | Non-<br>Randomized<br>Subjects | 16.2.7.1 | |
| | Listing | 16.2.7.3 | Incidents | All Randomized<br>Subjects | 16.2.7.3 | |
| 16.2.8 Oth | er Listings an | nd Listing of Labora | tory Measurements, when required by regulatory authors | orities (if applicable) | | |
| | Listing | 16.2.8.1 | Oral Soft Tissue Examination | All Randomized<br>Subjects | 16.2.8.1 | |





| CSR<br>Section | TLF | Number | Title | Population | Template | Topline |
|---|---|---|---|---|---|---|
| | Listing | 16.2.8.2 | Oral Hard Tissue Examination | All Randomized<br>Subjects | 16.2.8.2 | |
| 16.4 Individual Subject Data Listings | | | | | | |
| | NA | | | | | |